CLINICAL TRIAL: NCT05415735
Title: Total-Body PET Imaging to Understand the Physiology of Stress, Inflammation, and Meditation Following a Heart Attack
Brief Title: Stress Management and Resiliency Training Following Acute Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Michelle Dossett, Assistant Professor of Medicine, University of California, Davis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1787419
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Heart Attack; Cardiovascular Diseases
MeSH Terms: conditions — Myocardial Infarction; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMART Program (Experimental): The Stress Management and Resiliency Training (SMART) Program is a multimodal mind-body and cognitive skills-based program that teaches participants a variety of different approaches for reducing their physiologic stress response. The program is delivered virtually (online) for 1.5 hours once a week for 8 weeks.
  Interventions: Behavioral: Stress Management and Resiliency Training Program

INTERVENTIONS:
Behavioral: Stress Management and Resiliency Training Program — This is a multimodal mind-body program designed to teach participants a variety of different strategies to reduce their physiologic stress response.

SUMMARY:
The goal of this pilot study is to use total body PET/CT imaging to examine the relationships between stress, amygdala activation, and arterial wall inflammation in participants before and after participating in a multi-modal stress reduction program.

ELIGIBILITY:
Inclusion Criteria:

* Concurrently enrolled in an observational study of patients who have had an acute myocardial infarction
* Score on PSS-10 of 14 or greater during screening
* Willing and able to access the internet to participate in the online SMART Program

Exclusion Criteria:

* Poorly controlled physical or mental health condition that would likely interfere with the ability to participate in SMART or ability to undergo PET scan
* Current daily practice of meditation of 10 minutes or more per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Change in amygdala activation | about 10 weeks
  change in radiotracer uptake in the amygdala with FDG-PET imaging from before to after the SMART Program

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
Interested researchers need to submit a written request for access to data which will be reviewed internally. If approved, a data sharing agreement will need to be created.